CLINICAL TRIAL: NCT04270578
Title: German Study Gestational Diabetes (PREG)
Brief Title: Gestational Diabetes
Acronym: PREG
Status: Recruiting | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Deutsches Diabeteszentrum (DDZ), Leibniz-Institut Düsseldorf (Unknown); Medizinische Klinik und Poliklinik III, Universitätsklinikum Carl Gustav Carus, TU Dresden (Unknown); Klinik für Diabetologie an der Medizinischen Klinik - Innenstadt, LMU München (Unknown); Universitätsklinik Heidelberg, Abteilung Innere Medizin I, Schwerpunkt Endokrinologie und Stoffwechsel (Unknown); Universitätsklinikum Leipzig, IFB Adipositas Erkrankungen (Unknown)
Responsible Party: Sponsor
Other Study IDs: 218/2012BO2
Record Dates: First submitted 2019-11-15; First posted 2020-02-17 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Gestational Diabetes
Keywords: gestational diabetes; insulin
MeSH Terms: conditions — Diabetes, Gestational; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women with GDM
- Women without GDM

SUMMARY:
Due to a changed lifestyle with less physical activity, unfavorable diets rich in fat and calories and obesity, the prevalence of diabetes mellitus is increasing worldwide. The diabetes epidemic is associated with significant personal and socio-economic consequences. Despite attempts to prevent the complications of diabetes, this disease is still the leading cause of blindness, chronic renal insufficiency and non-traumatic amputation. It is important to detect early on an increase in blood sugar and treat it accordingly to reduce costs and to minimize the personal suffering of those affected. As the number of patients with type 2 diabetes mellitus continues to rise, the number of young women with gestational diabetes mellitus (GDM) also increases. This is a disorder og glucose metabolism, which occurs for the first time in pregnancy. The causes for this are manifold. Among other causes, the increasing age of the mothers and weight gain during pregnancy are risk factors for gestational diabetes. Although it has been recommended that women with gestational diabetes should be re-examined after the birth of their child, many women have not. The study is a follow-up study to clarify whether insulin secretion disorder in women with and after GDM is a risk factor for the occurrence of type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

- Signed and dated informed consent

Enrollment is possible during AND after gestation:

* Baseline visit (pregnancy): gestational week 24+0 till 31+6
* Postpartum visits: documented occurence of GDM in previous pregnancy

Exclusion Criteria:

* Age < 18years
* Diabetes Mellitus Type 1 or Type 2
* GFR < 60 ml/min/1,73 m2
* CRP > 1 mg/dl
* Increased levels of transaminases 2 fold above ULN
* Preexisting cardiac conditions
* Weight loss > 10% within 6 months prior to inclusion
* Psychiatric disorders
* Chronic alcohol or substance abuse
* Blood sugar increasing or decreasing drug therapy, e.g. steroids, antidiabetics, insulin
* only postpartum visits: pregnancy or lactation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women in gestational week 24+0 till 31+6 and women postpartum who had a documented occurence of GDM in previous pregnancy.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2012-05-23 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Glucose tolerance during 75 g oral glucose tolerance test | Glycemia from start of glucose tolerance test (0 minutes) until the end (120 minutes)
  Glucose tolerance, insulin sensitivity and insulin secretion during oral glucose tolerance test

SECONDARY OUTCOMES:
Glucose tolerance during 75 g oral glucose tolerance test 1, 2, 5, 10 years postpartum | Glycemia from start of glucose tolerance test (0 minutes) until the end (120 minutes)
  Glucose tolerance during oral glucose tolerance test
Body fat distribution | Once during pregnancy and 1, 2, 5, and 10 years postpartum
  Measurement of body fat distribution by MRS
Spiroergometry to assess physical fitness | 1, 2, 5, and 10 years postpartum
  Measurement of VO2max (l/min/kg) as a proxy for physical fitness
BIA (bioimpedance analysis) | Once during pregnancy and 1, 2, 5, and 10 years postpartum
  BIA to estimate body fat (%)
BMI | Once during pregnancy and 1, 2, 5, and 10 years postpartum
  Measurement of weight (kg) and height (m) and given as kg/m^2
Assessment of cognitive abilities in offspring | 6 and 10 years postpartum
  Cognitive skills represented as an intelligence quotient will be assessed Wechsler Intelligence Scale for Children - Fifth Edition (WISC-V)
Assessment of cognitive, motoric and language development in offspring | 2 years postpartum
  Cognitive, motoric and language development of children will be assessed with the Bayley Scales of Infant and Toddler Development - Third Edition (Bayley-III)
BIA in offspring | 2, 6 and 10 years postpartum
  BIA to estimate body composition in offspring
Electrocardiogram | 2, 6 and 10 years postpartum
  10 minute ECG to assess RR distance for calculation of heart rate variability (R wave distance in ms)
blood sample | 6 and 10 years postpartum
  blood sample to assess HbA1C

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Fritsche, MD, Principal Investigator — University Hospital Tuebingen
Locations (1):
- University Hospital Tuebingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bauer I, Schleger F, Hartkopf J, Veit R, Breuer M, Schneider N, Pauluschke-Frohlich J, Peter A, Preissl H, Fritsche A, Fritsche L. Pre-pregnancy BMI but not mild stress directly influences Interleukin-6 levels and insulin sensitivity during late pregnancy. Front Biosci (Landmark Ed). 2022 Feb 12;27(2):56. doi: 10.31083/j.fbl2702056. PMID 35226999
- [Derived] Fritsche L, Heni M, Eckstein SS, Hummel J, Schurmann A, Haring HU, Preissl H, Birkenfeld AL, Peter A, Fritsche A, Wagner R. Incretin Hypersecretion in Gestational Diabetes Mellitus. J Clin Endocrinol Metab. 2022 May 17;107(6):e2425-e2430. doi: 10.1210/clinem/dgac095. PMID 35180296
- [Derived] Fritsche L, Hummel J, Wagner R, Loffler D, Hartkopf J, Machann J, Hilberath J, Kantartzis K, Jakubowski P, Pauluschke-Frohlich J, Brucker S, Horber S, Haring HU, Roden M, Schurmann A, Solimena M, de Angelis MH, Peter A, Birkenfeld AL, Preissl H, Fritsche A, Heni M. The German Gestational Diabetes Study (PREG), a prospective multicentre cohort study: rationale, methodology and design. BMJ Open. 2022 Feb 15;12(2):e058268. doi: 10.1136/bmjopen-2021-058268. PMID 35168986